CLINICAL TRIAL: NCT02492009
Title: Patient Decision Aid (PDA) for Antidepressant Use In Pregnancy: a Pilot RCT
Brief Title: Patient Decision Aid for Antidepressant Use in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRAS project ID 166207; R&D2015/044 (Other: South London and Maudsley / IOP Office); REC reference 15/LO/0601 (Other: RES Committee London - Queen Square)
Record Dates: First submitted 2015-06-22; First posted 2015-07-08 (Estimated); Last update posted 2021-10-27 (Actual); Status verified 2016-09

CONDITIONS: Depression; Pregnancy
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Resource Sheet (Placebo Comparator): Women allocated to the control intervention will login to the study website and receive a printable PDF containing references to standard published information on antidepressant use in pregnancy. This ensures women have access to accurate information on the benefits and risks of antidepressant medication in pregnancy (even though they will not receive the PDA).
  Interventions: Behavioral: Standard Resource Sheet
- Electronic Patient Decision Aid (Active Comparator): The electronic Patient Decision Aid (PDA) is an interactive website with 3 main sections:
  1. Evidence-based information on (a) depression in pregnancy, (b) each treatment option and procedure;
  2. (a) Evidence-based information on the risks and benefits of both untreated depression and antidepressant treatment, (b) exercises to help women determine which risks and benefits are most important to them; and
  3. A summary section that outlines the information reviewed and which benefits and risks they deemed most important.
  At the end of the PDA, women allocated to this intervention will ALSO receive the standard resource sheet which is being used as the placebo comparator.
  Interventions: Behavioral: Patient Decision Aid

INTERVENTIONS:
Behavioral: Standard Resource Sheet — Women allocated to the control intervention will login to the study website and receive a printable PDF containing references to standard published information on antidepressant use in pregnancy. This ensures women have access to accurate information on the benefits and risks of antidepressant medication in pregnancy (even though they will not receive the PDA).
  Arms: Standard Resource Sheet
Behavioral: Patient Decision Aid — The electronic Patient Decision Aid (PDA) is an interactive website with 3 main sections:
  1. Evidence-based information on (a) depression in pregnancy, (b) each treatment option and procedure;
  2. (a) Evidence-based information on the risks and benefits of both untreated depression and antidepressant treatment, (b) exercises to help women determine which risks and benefits are most important to them; and
  3. A summary section that outlines the information reviewed and which benefits and risks they deemed most important.
  At the end of the PDA, women allocated to this intervention will ALSO receive the standard resource sheet which is being used as the placebo comparator.
  Arms: Electronic Patient Decision Aid

SUMMARY:
The proposed study is a pilot randomized controlled trial (RCT) of an electronic patient decision aid (PDA) for antidepressant use in pregnancy. The overall aim of this pilot RCT is to establish the feasibility of future large international RCT of the PDA's effectiveness.

DETAILED DESCRIPTION:
Depression in pregnancy is common, affecting up to 10% of women and represents serious risk to mother and infant. Unfortunately, antidepressant medication, a first-line treatment for depression in pregnancy, also comes with risks, making this a complex decision. Clinical care appears to be insufficient for ensuring that women make decisions that are consistent with their own values and with which they feel satisfied. Patient decision support tools can address such barriers. Canadian colleagues have created a patient decision aid (PDA) that has the potential to improve the decision-making process for women regarding antidepressant use in pregnancy in conjunction with clinical care. This study is a pilot RCT of the above PDA in London, to be conducted in parallel with a pilot RCT in Toronto.The overall objective of this project is to inform the development of a larger, international RCT to assess the efficacy of this PDA for antidepressant use in pregnancy. To achieve this objective, the investigators will assess the feasibility of the trial protocol to evaluate the PDA and determine the preliminary effect size for a larger multisite efficacy study. The primary outcome for this pilot study is the feasibility of conducting a large randomized controlled trial to evaluate the efficacy of the PDA. This includes feasibility (how well the trial protocol can be implemented), acceptability (usability and tolerability of the intervention) and adherence (the degree to which the trial protocol is followed). It is hypothesized that the protocol will be feasible, that the PDA will have a high degree of acceptability, and that adherence to the protocol will be high.

ELIGIBILITY:
INCLUSION CRITERIA: Women who meet all of the following criteria:

* Are aged over 18
* Are planning a pregnancy or are <30 weeks pregnant at enrolment
* Have been offered to start or continue an antidepressant as treatment for depression by their clinician a
* Have moderate-to-high decisional conflict (score of >25 on the Decisional Conflict Scale)

EXCLUSION CRITERIA: Women who meet any of the following criteria:

* Have had alcohol or drug abuse or dependence in the previous 12 months
* Have active suicidal ideation or psychosis
* Are incapable of consenting to participation
* Have any major obstetric complications or foetal cardiac anomaly in the current or in a past pregnancy,
* Are visually impaired
* Do not have sufficient English language proficiency to use the PDA.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Feasibility, measured by 'Recruitment Rate' | Up to one year from when the study starts enrolling participants

SECONDARY OUTCOMES:
Depression, measured by the Edinburgh Postnatal Depression Scale | (a) Baseline (pre-randomization) and (b) 4 Weeks post-randomization and (c) 12 weeks postpartum (for participants who enrolled while pregnant) OR 6 months post-randomization (for women who enrolled while planning a pregnancy)
Anxiety, measured by the Spielburg State-Trait Anxiety Inventory | (a) Baseline (pre-randomization) and (b) 4 Weeks post-randomization and (c) 12 weeks postpartum (for participants who enrolled while pregnant) OR 6 months post-randomization (for women who enrolled while planning a pregnancy)
Decisional conflict, measured by the Decisional Conflict Scale | Baseline (pre-randomization) and 4 Weeks post-randomization
Knowledge about antidepressant treatment in pregnancy | Baseline (pre-randomization) and 4 Weeks post-randomization
Intervention acceptability to patients, measured by the PDA Acceptability Questionnaire | 4 Weeks post-randomization]
Intervention acceptability to clinicians, measured by the Provider Perspective Survey | After follow-up data is complete (12 weeks postpartum if last patient was recruited in pregnancy, or 6 months after baseline interview if last patient was recruited when planning a pregnancy)
Treatment Decision(s) | (a) Baseline (pre-randomization) and (b) 4 Weeks post-randomization and (c) 12 weeks postpartum (for participants who enrolled while pregnant) OR 6 months post-randomization (for women who enrolled while planning a pregnancy)
Feasibility, measure by 'Time between recruitment to first log-in to the study website' | 4 weeks post-randomization
Feasibility, measured by 'Study Website Usage' | 4 Weeks post-randomization
  Composite measure comprised of: (1) number of participants who complete the PDA, (2)length of time required to complete the PDA, (3) number of log ins, (4) number of times the PDA is completed per participant, (5) total number of webpages viewed).
Feasibility, measured by 'Number of participants who follow-up with their physician during the intended timeline' | 4 weeks post-randomization
Feasibility, measured by 'The rate of follow-up data collection' | (a) 4 Weeks post-randomization and (b) 12 weeks postpartum (for participants who enrolled while pregnant) OR 6 months post-randomization (for women who enrolled while planning a pregnancy)

CONTACTS AND LOCATIONS:
Overall Officials: Louise M Howard, PhD, Principal Investigator — Section of Women's Mental Health, King's College London
Locations (1):
- South London and Maudsley NHS Foundation Trust, London, United Kingdom

REFERENCES:
- [Result] Khalifeh H, Molyneaux E, Brauer R, Vigod S, Howard LM. Patient decision aids for antidepressant use in pregnancy: a pilot randomised controlled trial in the UK. BJGP Open. 2019 Dec 10;3(4):bjgpopen19X101666. doi: 10.3399/bjgpopen19X101666. Online ahead of print. PMID 31822489
- See also: Related Info — https://bjgpopen.org/content/3/4/bjgpopen19X101666

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-01-22): https://cdn.clinicaltrials.gov/large-docs/09/NCT02492009/Prot_SAP_000.pdf
  • Informed Consent Form (2015-11-27): https://cdn.clinicaltrials.gov/large-docs/09/NCT02492009/ICF_001.pdf